CLINICAL TRIAL: NCT06487819
Title: Evaluation of Temporomandibular Joint Condition Post Longstanding Mouth Opening by Rubber Dam (A Clinical and Radiographic Study)
Brief Title: Evaluation of Temporomandibular Joint Condition Post Longstanding Mouth Opening by Rubber Dam
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, ‪Ahmed Sabry‬, Resident at Oral and Maxillofacial Surgery, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Screening
Other Study IDs: AUAREC202400002-16
Record Dates: First submitted 2024-06-19; First posted 2024-07-05 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Temporomandibular Joint Condition Post Longstanding Mouth Opening During Dental Procedure Using Rubber Dam; TMJ Disc Disorder; Osteoarthritis; Myofacial Pain
MeSH Terms: conditions — Osteoarthritis; Facial Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 - Short Duration Rubber Dam Application (Experimental): Patients undergoing dental procedures with rubber dam isolation for 30 to 60 minutes. This group will help assess the impact of short-term mouth opening on temporomandibular joint (TMJ) condition.
  Interventions: Procedure: Application of a rubber dam during dental treatments for varying durations.
- Group 2 - Medium Duration Rubber Dam Application (Experimental): Patients undergoing dental procedures with rubber dam isolation for 60 to 90 minutes. This group will help evaluate the effects of medium-term mouth opening on TMJ condition.
  Interventions: Procedure: Application of a rubber dam during dental treatments for varying durations.
- Group 3 - Long Duration Rubber Dam Application (Experimental): Patients undergoing dental procedures with rubber dam isolation for more than 90 minutes. This group will provide insights into the impact of long-term mouth opening on TMJ condition.
  Interventions: Procedure: Application of a rubber dam during dental treatments for varying durations.

INTERVENTIONS:
Procedure: Application of a rubber dam during dental treatments for varying durations. — Patients in each group will undergo dental procedures (either operative or endodontic treatment) with rubber dam isolation. The rubber dam will be applied for the specific durations mentioned in each group to evaluate the impact of mouth opening on the temporomandibular joint (TMJ).

SUMMARY:
This Clinical and radiographic study will be designed to evaluate the temporomandibular joint condition post longstanding mouth opening during dental procedure using rubber dam. primary outcome : preoperative and postoperative assessment of interincisal distance , occlusal biting force , visual analogue scale , lateral excursion movement and Magnetic resonance imaging (MRI).

Secondary outcome: investigator will try to answer the question of what is the best duration of time could the dentist use rubber dam isolation in dental procedures without harmful effect on TMJ and its supporting structures?

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged from 18 - 40 years old of both sexes.
2. No evidence of bad habits that affect occlusion like bruxism or clenching.
3. Patient with normal occlusion.
4. Patient free of any signs and symptoms of TMD and myofascial pain.
5. Normal range of TMJ movements.
6. Normal biting force.

Exclusion Criteria:

1. Patient with systemic or local diseases that can affect TMJ like osteoarthritis, rheumatoid arthritis, or systemic lupus erythema.
2. Patient with trismus.
3. Patient with Recurrent dislocation of TMJ.
4. Swelling affects mouth opening.
5. Patient came with TMJ ankylosis.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-08-10 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Interincisal Distance | Preoperative, immediately postoperative, 2 weeks postoperative.
  Measurement of the distance from the incisal edge of upper incisors to the incisal edge of lower incisors when the mouth is opened maximally in mm.
Occlusal Biting Force | Preoperative, immediately postoperative, 2 weeks postoperative.
  measurement of the biting force exerted by the patient's occlusion. This will be measured using a bite force gauge or similar instrument at the specified time points.
Visual Analogue Scale (VAS) | Preoperative, immediately postoperative, 2 weeks postoperative.
  A subjective measure of pain intensity experienced by the patient. Patients will mark their pain level on a scale from 0 (no pain) to 10 (worst pain imaginable).
Magnetic Resonance Imaging (MRI) | 2 weeks postoperative (for symptomatic patients).
  MRI scans will be done for patients who exhibit signs and symptoms of TMD postoperatively.
Lateral Excursion Movement | Preoperative, immediately postoperative, 2 weeks postoperative.
  The maximum amount of lateral excursion on each side will be measured in mm.

SECONDARY OUTCOMES:
Optimal Duration for Rubber Dam Use | immediately postoperative
  measure the duration of time for rubber dam application from the beginning of rubber dam application till the dentist remove rubber dam from the mouth of patient .

CONTACTS AND LOCATIONS:
Overall Officials: ‪Ahmed Sabry‬, Principal Investigator — Al-Azhar University
Locations (1):
- ‪Ahmed Sabry‬, Asyut, Assuit, Egypt

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Wang Q, Jia J, Zhou C, Ye W, Bi R. A Bibliometric Analysis of Research on Temporomandibular Joint Disc Displacement from 1992 to 2022. Healthcare (Basel). 2023 Jul 24;11(14):2108. doi: 10.3390/healthcare11142108. PMID 37510548
- [Background] Liu F, Steinkeler A. Epidemiology, diagnosis, and treatment of temporomandibular disorders. Dent Clin North Am. 2013 Jul;57(3):465-79. doi: 10.1016/j.cden.2013.04.006. PMID 23809304
- [Background] 3. Okeson JP. Management of Temporomandibular Disorders and Occlusion. 5th ed. Louis: Mosby; 2003.
- [Background] Goldstein BH. Temporomandibular disorders: a review of current understanding. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 1999 Oct;88(4):379-85. doi: 10.1016/s1079-2104(99)70048-x. PMID 10519741
- [Background] Huang GJ, Rue TC. Third-molar extraction as a risk factor for temporomandibular disorder. J Am Dent Assoc. 2006 Nov;137(11):1547-54. doi: 10.14219/jada.archive.2006.0090. PMID 17082281
- [Background] Sahebi S, Moazami F, Afsa M, Nabavi Zade MR. Effect of lengthy root canal therapy sessions on temporomandibular joint and masticatory muscles. J Dent Res Dent Clin Dent Prospects. 2010 Summer;4(3):95-7. doi: 10.5681/joddd.2010.024. Epub 2010 Sep 16. PMID 22991607
- [Background] Nasef M, Alashmawy M, Abdelrahman A, Elsaid M, Elwaseef S, Mohamed A. Evaluation of intra-articular injection of injectable platelet-rich fibrin, anterior repositioning splint and arthrocentesis in treatment of temporomandibular joint internal derangement. Br J Oral Maxillofac Surg. 2024 Oct;62(8):710-715. doi: 10.1016/j.bjoms.2024.05.002. Epub 2024 May 20. PMID 39043507
- [Background] Tiwari RVC, Managutti A, Lakshmi DP, Mohindru K, Damarasingu R, Dubey A. Isolation Systems and its Effectiveness in Oral and Maxillofacial Surgery: A Systematic Review. J Pharm Bioallied Sci. 2023 Jul;15(Suppl 1):S79-S85. doi: 10.4103/jpbs.jpbs_518_22. Epub 2023 Jul 5. PMID 37654409
- [Background] Cochran MA, Miller CH, Sheldrake MA. The efficacy of the rubber dam as a barrier to the spread of microorganisms during dental treatment. J Am Dent Assoc. 1989 Jul;119(1):141-4. doi: 10.14219/jada.archive.1989.0131. PMID 2760346